CLINICAL TRIAL: NCT01188694
Title: Enhancing Extinction Learning in Post Traumatic Stress Disorder (PTSD)
Acronym: HELP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Texas (Other); University of Pennsylvania (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lori Zoellner, Professor, Department of Psychology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 37340; R34MH087375 (NIH); 107654 (Other: FDA IND#)
Record Dates: First submitted 2010-07-20; First posted 2010-08-25 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-03

CONDITIONS: Chronic Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychotherapy; Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Psychotherapy plus Methylene Blue, USP (Experimental)
  Interventions: Drug: Psychotherapy plus Methylene Blue, USP
- Psychotherapy Plus Placebo (Placebo Comparator)
  Interventions: Behavioral: Psychotherapy plus Placebo
- Delayed Psychotherapy (Other)
  Interventions: Behavioral: Delayed Psychotherapy

INTERVENTIONS:
Drug: Psychotherapy plus Methylene Blue, USP — This treatment involves daily visits with a therapist for 50 to 60 minutes for a total of six sessions. At the end of each session, 260 mg of methylene blue, USP will be given.
  Arms: Psychotherapy plus Methylene Blue, USP
Behavioral: Psychotherapy plus Placebo — This treatment involves daily visits with a therapist for 50 to 60 minutes for a total of six sessions. At the end of each session, capsules containing the placebo will be given.
  Arms: Psychotherapy Plus Placebo
Behavioral: Delayed Psychotherapy — Individuals must wait approximately five to six weeks to start treatment. They will come in for two check-in appointments before starting treatment. Treatment will consist of ten twice-weekly psychotherapy sessions (90-120 min each session).
  Arms: Delayed Psychotherapy

SUMMARY:
Posttraumatic stress disorder (PTSD) is a condition that involves intense memories of a traumatic event and intense, persistent feelings of anxiety. There are several effective therapies for PTSD, but they are often time consuming. The investigators want to see if the investigators can shorten treatment time while keeping therapy effective by adding a medication called methylene blue, USP, taken orally as a pill, to the therapy. The specific aims are: 1) To see whether medication plus psychotherapy improves PTSD symptoms more than placebo plus psychotherapy or a waitlist; 2) To examine the long-term outcome of those receiving medication plus psychotherapy 1 and 3 months after treatment has ended; 3) To examine whether medication plus psychotherapy helps with depression, trauma-related cognitions, and functioning.

DETAILED DESCRIPTION:
The psychotherapy the investigators are offering in this study is a type of cognitive behavioral therapy called imaginal exposure. In imaginal exposure, the investigators encourage the client to approach the memory of the trauma by recounting the trauma story to the therapist and discussing his or her reactions to the memory.

ELIGIBILITY:
Inclusion Criteria:

1. Current primary PTSD diagnosis based on DSM-IV criteria, with a minimum duration of 12 weeks since the traumatic event.
2. Between the age of 18 and 65.

Exclusion Criteria:

1. Current diagnosis of schizophrenia, delusional disorder, or organic mental disorder as defined by the DSM-IV.
2. Current diagnosis of bipolar disorder, depression with psychotic features, or depression severe enough to require immediate psychiatric treatment (i.e., serious suicide risk with intent and plan).
3. Current diagnosis of alcohol or substance dependence within the 3 previous months.
4. Unwilling or unable to discontinue current trauma-focused psychotherapy or psychotropic medication (at least 1 month medication free).
5. Ongoing intimate relationship with the perpetrator (in assault-related PTSD cases).
6. Unstable cardiovascular, autoimmune, endocrine, neurological, renal, hepatic, retinal, gastrointestinal, or hematological disorder or current seizure disorder.
7. Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception for the duration of active treatment.
8. A history of hypersensitivity or allergy to MB.
9. Any condition possibly affecting drug absorption (e.g., gastrectomy).
10. Glucose-6-phosphate dehydrogenase deficiency.
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that, in the judgment of the Medical Directors, would make the participant inappropriate for entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Zoellner, PhD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas, Austin, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Zoellner LA, Telch M, Foa EB, Farach FJ, McLean CP, Gallop R, Bluett EJ, Cobb A, Gonzalez-Lima F. Enhancing Extinction Learning in Posttraumatic Stress Disorder With Brief Daily Imaginal Exposure and Methylene Blue: A Randomized Controlled Trial. J Clin Psychiatry. 2017 Jul;78(7):e782-e789. doi: 10.4088/JCP.16m10936. PMID 28686823

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psychotherapy Plus Methylene Blue, USP | Psychotherapy Plus Placebo | Delayed Psychotherapy
Started | 15 | 16 | 11
Completed | 10 | 15 | 10
Not Completed | 5 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psychotherapy Plus Methylene Blue, USP | Psychotherapy Plus Placebo | Delayed Psychotherapy | Total
Number analyzed (Participants) | 15 | 16 | 11 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 11 | 42
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 8 | 30
  Male | 5 | 4 | 3 | 12
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 11 | 42

OUTCOME MEASURES:

1. Primary Outcome: PTSD Symptom Severity-Interview (PSS-I)
Description: PTSD Symptom Scale - Interview Version, higher scores represent higher PTSD severity (range 0 - 51)
Time Frame: Pre-treatment, post-treatment (4 weeks from pre-), 1-month follow-up (from post-), and 3-month follow-ups (from post-)
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Psychotherapy Plus Methylene Blue, USP | Psychotherapy Plus Placebo | Delayed Psychotherapy
Number analyzed (Participants) | 15 | 16 | 11
units on a scale
  Pre-Treatment | 32.07 (6.17) | 31.38 (6.88) | 32.73 (7.24)
  Post-Treatment | 17.10 (10.57) | 14.67 (9.27) | 29.60 (8.40)
  1 Month Follow-up | 10.33 (3.77) | 13.33 (9.15) | 28.33 (7.43)
  3 Month Follow-up | 7.63 (5.53) | 10.93 (9.95) | 7.25 (9.82)

ADVERSE EVENTS:
Arm/Group | Psychotherapy Plus Methylene Blue, USP | Psychotherapy Plus Placebo | Delayed Psychotherapy
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/11
Other Adverse Events (participants affected / at risk) | 4/15 | 4/16 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Psychotherapy Plus Methylene Blue, USP (N=15) | Psychotherapy Plus Placebo (N=16) | Delayed Psychotherapy (N=11)
Nausea or Gastrointestinal (Gastrointestinal disorders) | 4 | 3 | 0
Anxiety or Depression (Psychiatric disorders) | 1 | 1 | 0
Eye Infection (Eye disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No